CLINICAL TRIAL: NCT05182073
Title: A Phase I Study of FT576 as Monotherapy and in Combination With Daratumumab in Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: FT576 in Subjects With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FT576-101
Record Dates: First submitted 2021-10-15; First posted 2022-01-10 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma; Myeloma
Keywords: Multiple Myeloma; daratumumab; CAR NK cell; cellular therapy; relapsed/refractory multiple myeloma; allogeneic natural killer cells; anti-CD38 monoclonal antibody; chimeric antigen receptor (CAR); BCMA; anti-B-cell maturation antigen (BCMA); natural killer (NK) cell
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Cyclophosphamide; fludarabine; daratumumab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Regimens A-A4 (Experimental): FT576 single dose monotherapy in subjects with r/r MM
  Interventions: Drug: FT576 (Allogenic CAR NK cells with BCMA expression); Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Bendamustine
- Regimen A1 (Experimental): FT576 multiple dose monotherapy in subjects with r/r MM
  Interventions: Drug: FT576 (Allogenic CAR NK cells with BCMA expression); Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Bendamustine
- Regimens B-B4 (Experimental): FT576 single dose in combination with daratumumab in subjects with r/r MM
  Interventions: Drug: FT576 (Allogenic CAR NK cells with BCMA expression); Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Daratumumab; Drug: Bendamustine
- Regimen B1 (Experimental): FT576 multiple dose in combination with daratumumab in subjects with r/r MM
  Interventions: Drug: FT576 (Allogenic CAR NK cells with BCMA expression); Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Daratumumab; Drug: Bendamustine

INTERVENTIONS:
Drug: FT576 (Allogenic CAR NK cells with BCMA expression) — Experimental Interventional Therapy: FT576 comprises allogeneic natural killer (NK) cells, derived from a clonal, CD38-knockout, human-induced pluripotent stem cell line (iPSC) that expresses anti-B-cell maturation antigen (BCMA) chimeric antigen receptor (CAR), high-affinity, non-cleavable CD16 (hnCD16), and IL-15/IL-15 receptor fusion protein (IL-15RF).
Drug: Cyclophosphamide — Conditioning Agent
Drug: Fludarabine — Conditioning Agent
Drug: Daratumumab — Anti-CD38 Monoclonal Antibody
  Other Names: Darzalex; Darzalex Faspro
  Arms: Regimen B1; Regimens B-B4
Drug: Bendamustine — Conditioning Agent
  Other Names: Bendeka; Treanda

SUMMARY:
This is a Phase I dose-finding study of FT576 as monotherapy and in combination with the monoclonal antibody daratumumab in multiple myeloma (MM). The study will consist of a dose-escalation stage and an expansion stage.

ELIGIBILITY:
* Abbreviated inclusion criteria:

Diagnosis of r/r MM with measurable disease by at least one of the following:

* Serum M-protein ≥1.0 g/dL
* Urine M-protein ≥200 mg/24 hours
* Involved serum free light chain level ≥10 mg/dL, with an abnormal kappa-lambda ratio if the serum M-protein <1.0 g/dL and/or urine M-protein <200 mg/24 hours
* Regimens A - A4 only: MM relapsed or progressed after ≥3 prior approved therapies, including an IMiD, proteosome inhibitor, and anti-CD38 mAb
* Regimens B - B4 only: MM relapsed or progressed after ≥2 prior approved therapies, including an IMiD and proteosome inhibitor

Note: for all Regimens, prior BCMA CAR T-cell therapy and BCMA-targeted therapy (e.g., bi-specific engagers or antibody-drug conjugates) is allowed

* Abbreviated exclusion criteria:

Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≥2

Evidence of insufficient hematologic function:

* ANC <1000/µL without growth factor support ≤7 days prior to measurement
* Platelet count <75,000/µL without platelet transfusion ≤72 hours prior to measurement

Evidence of insufficient organ function

* CrCL <50 ml/min by Cockcroft-Gault or other institutional method
* T bilirubin >1.5x ULN, except for Gilbert's syndrome
* AST >3x ULN or ALT >3x ULN, unless directly due to underlying malignancy
* O2 sat <92% on room air

Clinically significant cardiovascular disease:

* Myocardial infarction within 6 months of first treatment
* Unstable angina or CHF of NYHA Grade 2 or higher
* Cardiac EF <40%

Subjects with active central nervous system (CNS) , including leptomeningeal disease. Subjects with prior CNS involvement may be enrolled into the study if effective treatment of their CNS disease was completed at least 3 months prior to Day 1 with no evidence of disease clinically and at least stable findings on relevant CNS imaging.

Non-malignant CNS disease such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease or receipt of medications for these conditions in the 2-year period leading up to study enrollment

Currently receiving or likely to require immunosuppressive therapy (e.g., prednisone >5 mg daily) for any reason during the treatment period, with the exception of inhaled corticosteroids.

Clinically significant infections, including:

* HIV positive by serology
* HBV positive by serology or PCR
* HCV positive by serology or PCR

Live vaccine <6 weeks prior to start of conditioning

Receipt of an allograft organ transplant

Ongoing requirement for systemic graft -versus-host disease therapy

Plasma cell leukemia defined as a plasma cell count >2000/mm^3

Prior malignancy (other than current indication including any antecedent hematologic disorder) within the 2 years prior to enrollment except for the following: basal or squamous cell carcinomas of the skin, carcinoma in situ of the cervix or breast treated with curative intent, or localized prostate cancer treated with curative intent, or malignancy that, in the opinion of the investigator and Sponsor's Medical Monitor, is considered cured with minimal risk of recurrence within 3 years.

Washout periods from prior therapies:

- Chemotherapy, or radiation therapy, except for palliative purposes, within 14 days prior to the first dose of FT576 (Day 1) or five half-lives, whichever is shorter; Investigational therapy within 30 days prior to the first dose of FT576 study treatment or five half-lives, whichever is shorter; Biologic therapy (e.g., anti-CD38 mAbs or anti-SLAMF7 monoclonal antibodies), including autologous cellular immunotherapy (e.g. CAR-T/ CAR-NK), antibody-drug conjugates or bi-specific immune-cell engaging antibody within 30 days prior to first dose of FT576 (Day 1) or half -lives whichever is shorter. prior allogenic HSCT or allogenic CAR-T/CAR-NK within 6 months of first dose of FT576 (Day1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of DLTs within each dose-escalation cohort to determine the MTD or MAD | Cycle 1 Day -5 to Day 29 for Regimen A and A1; Cycle 1 Day -11 to Day 29 (each cycle is 40 days) for Regimen B and B1
Determine the RP2D which will be based on the overall safety and anti-tumor activity among the dose escalation and dose expansion cohorts | From FPI to LPI's end of Cycle 1 study treatment (End of cycle is Day 29 from Day 1 FT576 infusion)
Incidence, nature, and severity of adverse events | Cycle 1 Day -5 to Day 29 for Regimen A and A1; Cycle 1 Day -11 to Day 29 (each cycle is 40 days) for Regimen B and B1

SECONDARY OUTCOMES:
Objective response rate (ORR) | From baseline tumor assessment up to approximately 2 years after last dose of FT576
  Proportion of subjects with a best overall response of sCR, CR, VGPR, or PR, as determined by the investigator according to standard IMWG response criteria
Duration of response (DOR) | Up to 15 years
  Duration from the first occurrence of a documented objective response until the time of disease progression or relapse, or death due to progressive disease, as determined by the investigator according to standard IMWG response criteria
Progression-free survival (PFS) | Up to 15 years
  Time from first dose of study treatment to disease progression or relapse, or to the day of death from any cause, as determined by the investigator according to standard IMWG response criteria
Relapse-free survival (RFS) from complete response (CR) | Up to 15 years
  Duration from the start of sCR or CR until the time of relapse from sCR or CR, as determined by the investigator according to standard IMWG response criteria
Overall survival (OS) | Up to 15 years
  Time from first dose of study treatment to death from any cause
Pharmacokinetics (PK) of FT576 | From Baseline to PTFU visit of last cycle on the study treatment (End of cycle is Day 29 from Day 1 FT576 infusion of this cycle)
  Concentration of FT576 in peripheral blood following FT576 administration

CONTACTS AND LOCATIONS:
Overall Officials: Fate Trial Disclosure, Study Director — Fate Therapeutics, Inc
Locations (14):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope, Duarte, California
  - Scri-Cbci, Denver, Colorado
  - Medical Oncology Hematology Consultants, Newark, Delaware
  - Indiana University, Indianapolis, Indiana
  - University of Minnesota, Saint Paul, Minnesota
  - Washington University, St Louis, Missouri
  - Roswell Park, Buffalo, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Oncology Hematology Care, Inc, Cincinnati, Ohio
  - Tennessee Oncology - Nashville, Nashville, Tennessee
  - Texas Oncology-Medical City Dallas, Dallas, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ASH Dec 2020 Abstract — https://ash.confex.com/ash/2020/webprogram/Paper142750.html